

# STATISTICAL ANALYSIS PLAN

A Phase 2 Multi-Center, Randomized, Double Masked, Placebo Controlled Study to Assess the Safety and Efficacy of ST-100 Ophthalmic Solution in Subjects Diagnosed with Dry Eye Disease

Sponsor: Stuart Therapeutics, Inc.

411 SE Osceola St., Suite 203

Stuart, FL 34994 USA

Protocol Number: ST100-001

Author:



Date: 250CT2021

Version: 1.0



A Phase 2 Multi-Center, Randomized, Double Masked, Placebo Controlled Study to Assess the Safety and Efficacy of ST-100 Ophthalmic Solution in Subjects Diagnosed with Dry Eye Disease

Protocol Number: ST100-001

SAP Version: 1.0

**SAP Date:** 25OCT2021





A Phase 2 Multi-Center, Randomized, Double Masked, Placebo Controlled Study to Assess the Safety and Efficacy of ST-100 Ophthalmic Solution in Subjects Diagnosed with Dry Eye Disease

Protocol Number: ST100-001

SAP Version: 1.0

SAP Date: 25OCT2021

**Statistical Analysis Plan Approval** 





## **Document History**

SignNow E-Signature Audit Log

All dates expressed in MM/DD/YYYY (US)

**Document name:** Stuart Therapeutics Inc ST100-001 SAP draft v1.0 25-OCT-2021 clean

**Document created:** 10/26/2021 14:28:35

Document pages: 48

**Document ID:** 2fce7f547f0b437bad5cd8831715c2c12a6b22a2

**Document Sent:** 10/26/2021 14:31:54 UTC

Document Status: Signed

10/29/2021 17:36:43UTC





## **Table of Contents**

| 1. | Introduction | 8 |
|---|---|---|
| 2. | Study Objectives | 8 |
| 3. | Study Variables | 8 |
| 3.1 | Primary Endpoints | 8 |
| 3.2 | Secondary Endpoints | 8 |
| 3.3 | Safety Variables | 9 |
| 3.4 | Statistical Hypotheses | 9 |
| 3.5 | Estimands | 10 |
| 4. | Study Design and Procedures | 11 |
| 4.1 | General Study Design | 11 |
| 4.2 | Schedule of Visits and Assessments | 11 |
| 5. | Study Treatments | 12 |
| 5.1 | Method of Assigning Subjects to Treatment C | Groups12 |
| 5.2 | Masking and Unmasking | 12 |
| 6. | Sample Size and Power Considerations | 13 |
| 7. | Data Preparation | 13 |
| 7.1 | Input Data | 13 |
| 7.2 | Output Data | 13 |
| 8. | Analysis Populations | 14 |
| 8.1 | Intent-to-Treat | 14 |
| 8.2 | Per Protocol | 14 |
| 8.3 | Safety | 14 |
| 9. | General Statistical Considerations | 14 |
| 9.1 | Unit of Analysis | 14 |
| 9.2 | Missing or Inconclusive Data Handling | 14 |
| 9.3 | Definition of Baseline | 16 |
| 9.4 | Data Analysis Conventions | 16 |
| 9.5 | Adjustments for Multiplicity | 16 |
| 10. | Disposition of Subjects | 17 |
| 11. | Demographic and Pretreatment Variables | 18 |
| 11.1 | Demographic Variables | 18 |
| 11.2 | Baseline Disease Characteristics | 18 |
| 12. | Medical History and Concomitant Medication | s19 |
| 12.1 | Medical History | 19 |
| 12.2<br>25OC | | 19<br>& Proprietary Page 3 o |



| 12.3 Conco | mitant Procedures | 20 |
|---|---|---|
| 13. Dosing | g Compliance and Treatment Exposure | 20 |
| 13.1 Dosing | g Compliance | 20 |
| 13.2 Treatn | nent Exposure | 21 |
| 14. Efficad | cy Analyses | 21 |
| 14.1 Prima | ry Analysis | 21 |
| 14.1.1. | , , | 22<br>22 |
| 14.1.1.<br>14.1.1. | 1 1 07 | |
| 14.1.1. | , , | |
| 14.1.2.<br>14.1.2.<br>14.1.2. | 2 Multiple Imputation Methodology | 26<br>26<br>26<br>28 |
| 14.1.2. | 4 Figuresdary Analyses | |
| 14.2.3 | Analysis of Secondary Endpoints | |
| 14.2.1 | Corneal and Conjunctival Fluorescein staining (Ora Calibra® scale) | |
| 14.2.2 | Corneal and Conjunctival Lissamine Green staining (Ora Calibra® scale) | |
| 14.2.3 | Tear Film Break-Up Time | |
| 14.2.4 | · | |
| | Conjunctival Redness (Ora Calibra Scale) | |
| 14.2.6 | Drop Comfort Assessment | |
| 14.2.7 | Ocular Surface Disease Index | |
| 14.2.8 | Overall Ocular Discomfort & 4-Symptom Questionnaire (Ora Calibra® Scale). | |
| 14.2.9<br>14.2.9.<br>14.2.9. | | 33 |
| 14.2.10 | Visual Analog Scale | 33 |
| 14.2.11 | Unanesthetized Schirmer's Test | 33 |
| 15. Summ | ary of Efficacy Analyses | 34 |
| 16. Safety | Analyses | 34 |
| 16.1 Advers | se Events | 34 |
| 16.2 Best-0 | Corrected Visual Acuity (Early Treatment Diabetic Retinopathy Study) | 36 |
| 16.3 Slit-La | mp Biomicroscopy Examination | 36 |
| 16.4 Intraod | cular Pressure | 37 |
| 16.5 Undila | ted Fundoscopy Examination | 37 |
| | Pregnancy Test | |



| 17. | Interim Analyses | 37 |
|-----|---------------------------------------------------|----|
| 18. | Changes from Protocol-Stated Analyses | 37 |
| 19. | References | 37 |
| | Revision History | |
| 21. | Tables | 38 |
| 22. | Listings | 41 |
| 23. | Figures | 43 |
| 24. | Appendices | 44 |
| 24. | 1 Appendix 1: Schedule of Visits and Measurements | 44 |



## **List of Abbreviations**

| ADaM | Analysis Data Model |
|-----------|-----------------------------------------------|
| AE | Adverse Event |
| ANCOVA | Analysis of Covariance |
| ATC | Anatomical Therapeutic Chemical |
| BCVA | Best-Corrected Visual Acuity |
| BID | Bis in die (Twice Daily) |
| CAE® | Controlled Adverse Environment |
| CFB | Change from Baseline |
| CFV2-Post | Change from Visit 2 (Day 1) Post-CAE® |
| CI | Confidence Interval |
| CRO | Contract Research Organization |
| CS | Clinically Significant |
| DED | Dry Eye Disease |
| eCRF | Electronic Case Report Form |
| EDC | Electronic Data Capture |
| ETDRS | Early Treatment of Diabetic Retinopathy Study |
| IB | Investigator's Brochure |
| ICH | International Conference on Harmonisation |
| IOP | Intraocular Pressure |
| IP | Investigational Product |
| ITT | Intent-to-Treat |
| IWRS | Interactive Web Response System |
| LOCF | Last Observation Carried Forward |
| logMAR | Logarithm of the Minimum Angle of Resolution |
| LS | Least Squares |
| MCMC | Markov Chain Monte Carlo |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NCS | Not Clinically Significant |
| OD | Oculus dexter (Right Eye) |
| OS | Oculus sinister (Left Eye) |
| PDF | Portable Document Format |
| PMM | Pattern Mixture Model |
| PP | Per Protocol |
| PT | Preferred Term |
| RTF | Rich Text Format |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SDC | Statistics & Data Corporation |
| SDTM | Study Data Tabulation Model |
| SE | Standard Error |



| SOC | SOC System Organ Class |
|---|---|
| TEAE Treatment-Emergent Adverse Event | |
| TFBUT Tear Film Break-Up Time | |
| TMF Trial Master File | |
| WHODrug World Health Organization Drug Dictionary | |



#### 1. Introduction

The purpose of this statistical analysis plan (SAP) is to describe the planned analyses and reporting for protocol amendment 1 dated 21-MAY-2021.

This SAP is being written with due consideration of the recommendations outlined in the most recent International Conference on Harmonisation (ICH) E9 Guideline entitled Guidance for Industry: Statistical Principles for Clinical Trials, the most recent ICH E9 (R1) Guideline entitled Guidance for Industry: Statistical Principles for Clinical Trials: Addendum: Estimands and Sensitivity Analysis in Clinical Trials, and the most recent ICH E3 Guideline entitled Guidance for Industry: Structure and Content of Clinical Study Reports.

This SAP describes the data that will be analyzed and the subject characteristics, efficacy, and safety assessments that will be evaluated. This SAP provides details of the specific statistical methods that will be used. The statistical analysis methods presented in this document will supersede the statistical analysis methods described in the clinical protocol. If additional analyses are required to supplement the planned analyses described in this SAP, they may be completed and will be identified in the clinical study report.

#### 2. Study Objectives

The objective of this study is to compare the safety and efficacy of two different concentrations of ST-100 Ophthalmic Solution to placebo for the treatment of the signs and symptoms of dry eye.

#### 3. Study Variables

#### 3.1 Primary Endpoints

The primary efficacy endpoints are the following:

- Sign: Total corneal fluorescein staining score on the Ora Calibra® scale, measured by
- Symptom: Ocular discomfort score on the Ora Calibra® Ocular Discomfort Scale, measured by

#### 3.2 Secondary Endpoints

The secondary efficacy endpoints include the following:

- Fluorescein staining (Ora Calibra® scale) at Visits 3, 4, 5, 6, and 7 (Pre-CAE®, Post-CAE®, and Pre-to Post-CAE®): regions:
- Lissamine green staining (Ora Calibra<sup>®</sup> scale) at Visits 3, 4, 5, 6, and 7 (Pre-CAE<sup>®</sup>, Post-CAE<sup>®</sup>, and Pre- to Post-CAE<sup>®</sup>): regions:



- Tear film break-up time (TFBUT) at Visits 3, 4, 5, 6, and 7 (Pre-CAE<sup>®</sup>, Post-CAE<sup>®</sup>, and Pre- to Post-CAE<sup>®</sup>)
- Conjunctival Redness at Visits 3, 4, 5, 6, and 7 (Pre-CAE<sup>®</sup>, Post-CAE<sup>®</sup>, and Pre- to Post-CAE<sup>®</sup>)
- Drop comfort assessment after randomization at Visit 2 and Visit 6
- Ocular Surface Disease Index (OSDI<sup>®</sup>) at Visits 3, 4, 5, 6, and 7 (Pre-CAE<sup>®</sup>)
- Overall Ocular Discomfort and Four-symptom Questionnaire at Visits 3, 4, 5, 6, and 7 (Pre-CAE<sup>®</sup>, Post-CAE<sup>®</sup>, and Pre- to Post-CAE<sup>®</sup>)
- Ocular discomfort during CAE<sup>®</sup> at Visits 5, 6, and 7
- Daily diary
- Visual Analog Scale Burning/Stinging, Itching, Foreign Body Sensation, Blurred Vision, Eye Dryness, Photophobia, and Pain at Visits 3, 4, 5, 6, and 7 (Pre-CAE<sup>®</sup>)
- Unanesthetized Schirmer's Test at Visit 7 (Pre-CAE®)
- Ocular Discomfort Scale outside of the CAE<sup>®</sup> at Visits 3, 4, 5, 6, and 7 (Pre-CAE<sup>®</sup>, Post-CAE<sup>®</sup>, and Pre- to Post-CAE<sup>®</sup>)

#### 3.3 Safety Variables

The safety variables include the following:

- Best-corrected visual acuity (BCVA)
- Slit-lamp evaluation
- Adverse event (AE) query
- Intraocular pressure (IOP)
- Undilated fundoscopy

#### 3.4 Statistical Hypotheses







#### 3.5 Estimands

The primary comparisons in this trial will be between ST-100 Ophthalmic Solution (high dose or low dose) versus placebo at Day 29 in the Intent-to-Treat (ITT) population with multiple imputation using the following primary estimand:

#### Estimand 1:

Population:

Endpoint:

Intercurrent event:





## 4. Study Design and Procedures

#### 4.1 General Study Design

Study visits will be referred to in all tables and listings as the visit number and expected study day corresponding to the visit to enable reviewers to understand the assessment timing without referring to the protocol visit schedule. Table 1 shows the scheduled study visits, their planned study day (note: that there is no Day 0 and that Day 1 corresponds to the day of randomization), and the acceptable visit window for each study visit:

**Table 1. Study Visit Windows** 

| Scheduled Visit | Planned Study Day | Visit Window |
|-----------------|-------------------|--------------|
| Visit 1 | Day -7 | ± 1 day |
| Visit 2 | Day 1 | N/A |
| Visit 3 | Day 2 | ± 2 hours |
| Visit 4 | Day 4 | ± 2 hours |
| Visit 5 | Day 8 | ± 1 day |
| Visit 6 | Day 15 | ± 1 day |
| Visit 7 | Day 29 | ± 2 days |

## 4.2 Schedule of Visits and Assessments

The schedule of visits and assessments is provided in Appendix 1.



## 5. Study Treatments

#### 5.1 Method of Assigning Subjects to Treatment Groups

Before the initiation of study run-in at Visit 1 (Day -7), each subject who provides written informed consent will be assigned a screening number. All screening numbers will be assigned in strict numerical sequence at a site and no numbers will skipped or omitted. Each subject who meets all the inclusion and none of the exclusion criteria at Visit 1 (Day -7) and Visit 2 (Day 1) will be assigned a randomization number at the end of Visit 2 (Day 1). The Interactive Web Response System (IWRS) will be used to assign all randomization numbers.

Subjects will be randomized to one of the following treatment arms at Visit 2 (Day 1):

- Low dose ST-100 Ophthalmic Solution:
  High dose ST-100 Ophthalmic Solution:
- Placebo Ophthalmic Solution (Vehicle):

Approximately subjects will be randomly assigned to one of the three groups (1:1:1) to receive either ST-100 Ophthalmic Solution or placebo solution as topical ophthalmic drops administered bilaterally BID for 4 weeks. Subjects, Sponsor, Contract Research Organization (CRO), and site personnel will be masked to treatment assignment. Randomization and kit numbers will be assigned automatically to each subject as they are entered into the IWRS.

The site staff will dispense kit(s) required until the next visit. Both the randomization number and the dispensed study drug kit number(s) will be recorded on the subject's source document and electronic case report form (eCRF). Subjects, Sponsor, CRO, and site personnel will be masked to treatment assignment.

#### 5.2 Masking and Unmasking

All subjects, investigators, and study personnel involved with the conduct of the study will be masked with regard to treatment assignments. When medically necessary, the investigator may need to determine what treatment group has been assigned to a subject. When possible (i.e., in non-emergent situations), Ora and/or the study sponsor should be notified before unmasking study drug. Ora and/or the study Sponsor must be informed immediately about any unmasking event.

If an investigator identifies a medical need for unmasking the treatment assignment of a subject, he/she should contact Ora and/or the medical monitor prior to unmasking the identity of the investigational product (IP), if possible. Ora will ask the site to complete and send them the Unmasking Request Form. Ora will notify the Sponsor and jointly will determine if the unmasking request should be granted. They may consult the medical monitor as needed. The result of the request will be documented on the Unmasking Request Form. If approval is granted to unmask a subject, written permission via the Unmasking Request Form will be provided to the investigator. The investigator will unmask the subject using IWRS. The investigator will



complete the Unmasking Memo form and include it in the subject's study file and provide a copy for the Trial Master File (TMF). For each unmasked request, the reason, date, signature, and name of the person who unmasked the subject must be noted in the subject's study file.

Unmasked subjects will be discontinued from the study. Unmasked subjects will be followed for safety monitoring until resolution of the AE or study completion, whichever occurs last.

#### 6. Sample Size and Power Considerations

This study is expected to enroll subjects in each group, for a total of randomized subjects. Approximately subjects will be screened. Assuming a 10% drop out rate, subjects per group are expected to complete the study.

#### 7. Data Preparation

#### 7.1 Input Data

Study data will primarily be recorded on the eCRFs supplied by Statistics & Data Corporation (SDC) using iMedNet v1.211.1.

When all prerequisites for database lock have been met, the database will be locked. Following database lock, approval will be obtained from the Sponsor to unmask the study. Any changes to the database after data have been locked can only be made with the approval of the Sponsor in consultation with SDC.

Final analysis will be carried out after the following have occurred:

- Database lock has occurred with written authorization provided by appropriate SDC and Sponsor personnel.
- Protocol deviations have been identified and status defined (major/minor deviations) prior to database lock.
- Analysis populations have been determined.
- Randomized treatment codes have been unmasked.

#### 7.2 Output Data

Data from electronic data capture (EDC) and external data will be transferred to Biostatistics and incorporated into standard formats following the Study Data Tabulation Model (SDTM). Data will then be mapped to analysis datasets using the Analysis Data Model (ADaM). Both SDTM- and ADaM-formatted data will be used to create the subject listings, while all tables and figures will be based on the ADaM-formatted data.

SDTM will follow the SDTM version 1.7 model and will be implemented using the SDTM Implementation Guide version 3.3, and the most recent version of SDTM Controlled Terminology at the start of the study. ADaM data will follow the ADaM version 2.1 model and will be implemented using the ADaM



Implementation Guide version 1.2. Both SDTM and ADaM will be validated using Pinnacle 21 version 3.1.2. Any discrepancies in the validation will be noted in reviewer's guides accompanying the final data transfers.

Define.xml will be created for SDTM and ADaM using the Define-XML version 2.0 model.

| 8.1 Intent-to-Treat |
|---|
| The intent-to-treat (ITT) population includes |
| 8.2 Per Protocol |
| The per protocol (PP) population includes |
| 8.3 Safety |
| The safety population includes |
| The salety population includes |
| 9. General Statistical Considerations |
| 9.1 Unit of Analysis |
| Safety endpoints will be analyzed for both eyes. For efficacy endpoints, the unit of analysis will be the study |
| eye, or the "worst eye," as defined by the following: |
| Study (Worst) Eye: |

## 9.2 Missing or Inconclusive Data Handling

Imputation of missing data will be executed for partial or missing dates where complete dates are required to flag data as treatment-emergent or concomitant with treatment. Partial/missing start and end dates for AEs and concomitant medications will be imputed as follows:

Partial/missing start date:



- Dates with missing day only will be imputed as the 1st of the month unless the month and year are same as the month and year of first dose of study medication, in which case missing day will be imputed as the first dose day of study medication.
- Dates with both day and month missing will be imputed as 1 Jan unless the year is same as the
  year of first dose of study medication, in which case missing day and month will be imputed as the
  first dose day and month of study medication.
- Completely missing dates will be imputed as the first dose date of study medication unless the end date is on or before the first dose date of study medication, in which case missing date will be imputed as 1 Jan of the same year as the end date.

#### Partial/missing end date:

- Dates with missing day only will be imputed as the last day of the month unless the month and year
  are the same as the month and year of the last dose of study medication, in which case missing
  day will be imputed as the last dose day of study medication.
- Dates with both day and month missing will be imputed as 31 Dec unless the year is same as the
  year of the last dose of study medication, in which case missing day and month will be imputed as
  the last dose day and month of study medication.
- If the ongoing flag is missing or "Yes" then the date will not be imputed unless death date is available, in which case the missing date will be imputed as the death date. If ongoing is "No" then the missing end date will be imputed as the last dose date.
- If the imputed date is after the date of death, then the end date will be set equal to the date of death.

The original dates will be displayed in data listings and the imputed dates will be used in derivations only (study day, treatment-emergence status, etc).

Missing data for the primary efficacy endpoints will be imputed using multiple imputation on the ITT population as specified in Estimand 1 for primary analyses.

Sensitivity analyses of the primary efficacy analyses will include the following in order to provide a robust understanding of the impact of missing and spurious data:





#### 9.3 Definition of Baseline



#### 9.4 Data Analysis Conventions

All data analysis will be performed by SDC after the study is completed and the database has been locked and released for unmasking. Statistical programming and analyses will be performed using SAS® version 9.4 or higher. Output will be provided in rich text format (RTF) for tables and portable document format (PDF) for tables, listings, and figures using landscape orientation. All study data will be listed by subject, treatment, and visit (as applicable) based on all randomized subjects unless otherwise specified.

Summaries for continuous and ordinal variables will include the number of observations (n), arithmetic mean, standard deviation (SD), median, minimum, and maximum. Minima and maxima will be reported with the same precision as the raw values; means and medians will be presented to one additional decimal place than reported in the raw values. Standard deviations will be presented to two additional decimal places than reported in the raw values. Summaries for discrete variables will include counts and percentages. All percentages will be rounded to one decimal place (i.e., XX.X%). Differences between active treatment groups and placebo will be calculated as active minus placebo and change from baseline will be calculated as follow-up visit minus baseline.



Unless otherwise specified, summaries will be presented by treatment group and, where appropriate, visit. Listings will be sorted by treatment group, subject number, visit/time point, and parameter as applicable.

#### 9.5 Adjustments for Multiplicity







#### 10. Disposition of Subjects

Subject disposition will be presented in terms of the numbers and percentages of subjects who were included in the following analysis populations:

Subjects who are not discontinued from the study will be considered study completers. Disposition will be summarized by

The total number of screened subjects with the number and percentage of screen failure subjects.

The reasons for premature study discontinuation will be summarized by treatment group for all discontinued subjects. Percentages will be calculated using discontinued subjects as the denominator. The reasons for study discontinuation that will be summarized include: AE, protocol violation, administrative reasons, sponsor termination of study, subject choice, lost to follow-up, lack of efficacy, and other. The subset of COVID-19-related discontinuations will be summarized as well. A subject listing will be provided that includes the date of and reason for premature study discontinuation. The listing will indicate COVID-19 relatedness with a reason for COVID-19 relatedness.





| <u> </u> | | | |
|----------|---|---|---|
| | • | · | · |

For all screen failures, the reasons for screen failure will be displayed with the percentages calculated using total number of screen failures as the denominator.

In addition, subject listings will be provided that include informed consent date, screen failure reason, and exclusions from analysis populations. Details of the study randomization, including randomization date and time, randomized treatment, and actual treatment, will also be included within a subject listing. A listing summarizing all COVID-19-related discontinuations and protocol deviations will be generated as well.

#### 11. Demographic and Pretreatment Variables

#### 11.1 Demographic Variables

The demographic variables collected in this study include age, sex, childbearing potential for female subjects, race, ethnicity, and iris color. Subjects who record more than one race will be grouped into a single category denoted as Multiple. Iris color will be summarized at the eye level (OD and OS). Demographic variables will be summarized for the ITT and Safety populations, separately.

Age (years) will be summarized, overall and by treatment, using continuous descriptive statistics. Age will also be categorized as follows:

Age will be reported in years and calculated using the following formula:

The number and percentage of subjects will be presented, overall and by treatment, for age category, sex, race, ethnicity, and iris color.

A subject listing that includes all demographic variables will be provided for all screened subjects.

#### 11.2 Baseline Disease Characteristics

Baseline disease characteristics will be summarized by treatment group using



| 40 | Medical History and Concomitant Medications |
|----|---------------------------------------------|

#### 12.1 **Medical History**

Medical history will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) 24.0.



Listings of medical history will be generated separately for ocular and non-ocular data.

#### 12.2 **Concomitant Medications**

Concomitant medications will be coded using World Health Organization Drug Dictionary (WHODrug) Global (B3, March 2021) and summarized to the therapeutic drug class (Anatomical Therapeutic Chemical [ATC] 4 classification) and preferred name. If the ATC 4 classification is not provided, then the next lowest classification that is provided in the coding dictionary will be used. The preferred name will be defined as the active ingredient; if the active ingredient is not provided or includes more than two ingredients (e.g., multivitamins), then the drug name will be summarized as the preferred name. Any uncoded terms will be summarized under the ATC classification and preferred name of "Uncoded."

Concomitant medications are defined as those medications listed as having been taken (1) prior to initiation of randomized study drug administration and continuing for any period of time following the first administration of randomized study drug or (2) at any time following the first administration of randomized study drug. Prior medications are defined as those listed as having been prior to initiation of randomized study drug administration but not taken for any instance following the first administration of randomized study drug.





Listings of concomitant medications will be generated separately for ocular and non-ocular data.

#### 12.3 Concomitant Procedures

Concomitant procedures will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) 24.0.

Listings of concomitant procedures will be generated separately for ocular and non-ocular data.

#### 13. Dosing Compliance and Treatment Exposure

#### 13.1 Dosing Compliance

Dosing compliance (% compliance) will be assessed by calculating the number of actual doses received and comparing that to the number of expected doses as follows:



The number of actual doses received will be calculated from the number of used ampules from the study drug accountability eCRF. The number of expected doses that will be used for calculating compliance will be calculated as:



subjects that are lost to follow-up will be calculated as:

The number of expected doses for subjects who discontinue on visit 2 will be 2 doses.

A categorical dosing compliance variable will also be derived as non-compliant and over compliant

Dosing compliance (%) will be summarized with continuous descriptive statistics for each treatment group using the Safety population. The compliance category defined above will be summarized with discrete summary statistics.



A subject listing of dosing compliance will also be produced. In addition, the following listings will be produced for all randomized subjects:

- run-in and study drug assignment, dispensation, replacement, and study drug instillation;
- study drug accountability;

#### 13.2 Treatment Exposure

Extent of treatment exposure for completed or discontinued subjects will be calculated in days using the following:



Extent of treatment exposure for subjects who were lost to follow-up will be calculated in days using the following:

The extent of treatment exposure for subjects who discontinue on Visit 2 (Day 1) will be 1 day.

Extent of treatment exposure for each subject exposed to study drug will be summarized with continuous

descriptive statistics for each treatment group using the Safety population. Total exposure in days will be summarized for each treatment group as well. A subject listing of treatment exposure will also be produced.

#### 14. Efficacy Analyses

#### 14.1 Primary Analysis

The primary efficacy endpoints are the following:





# 14.1.1 Change from Baseline of Total Corneal Fluorescein Staining (Ora Calibra® Scale) in the Study Eye at Visit 7 (Day 29) Pre-CAE®





## 14.1.1.2 MULTIPLE IMPUTATION METHODOLOGY



























#### 14.1.2.3 ADDITIONAL SENSITIVITY ANALYSES

Additional sensitivity analyses will be conducted as described in <u>Section 14.1.1.3</u>.

#### 14.1.2.4 FIGURES



#### 14.2 Secondary Analyses

The secondary efficacy variables include the following:

- Fluorescein staining (Ora Calibra<sup>®</sup> scale) at Visits 3, 4, 5, 6, and 7 (Pre-CAE<sup>®</sup>, Post-CAE<sup>®</sup>, and Change from Pre-CAE<sup>®</sup> to Post-CAE<sup>®</sup>): regions:
- Lissamine green staining (Ora Calibra® scale) at Visits 3, 4, 5, 6, and 7 (Pre-CAE®, Post-CAE®, and Pre- to Post-CAE®): regions:
- TFBUT at Visits 3, 4, 5, 6, and 7 (Pre-CAE®, Post-CAE®, and Change from Pre-CAE® to Post-CAE®)
- Conjunctival Redness at Visits 3, 4, 5, 6, and 7 (Pre-CAE<sup>®</sup>, Post-CAE<sup>®</sup>, and Change from Pre-CAE<sup>®</sup> to Post-CAE<sup>®</sup>)
- Drop comfort assessment after randomization at Visit 2 and Visit 6
- OSDI<sup>©</sup> at Visits 3, 4, 5, 6, and 7 (Pre-CAE<sup>®</sup>)
- Four symptom questionnaire at Visits 3, 4, 5, 6, and 7 (Pre-CAE®, Post-CAE®, and Change from Pre-CAE® to Post-CAE®)
- Ocular discomfort during CAE<sup>®</sup> at Visits 5, 6, and 7
- Daily diary
- Visual Analog Scale Burning/Stinging, Itching, Foreign Body Sensation, Blurred Vision, Eye Dryness, Photophobia, and Pain at Visits 3, 4, 5, 6, and 7 (Pre-CAE®)



- Unanesthetized Schirmer's Test at Visit 7 (Pre-CAE®)
- Ocular Discomfort Scale outside of the CAE® at Visits 3, 4, 5, 6, and 7 (Pre-CAE®, Post-CAE®, and Change from Pre-CAE® to Post-CAE®)

#### 14.2.1 ANALYSIS OF SECONDARY ENDPOINTS



Subject listings will be provided for all efficacy endpoint assessments for randomized subjects only.



# 14.2.2 CORNEAL AND CONJUNCTIVAL FLUORESCEIN STAINING (ORA CALIBRA® SCALE) 14.2.3 CORNEAL AND CONJUNCTIVAL LISSAMINE GREEN STAINING (ORA CALIBRA® SCALE) 14.2.4 TEAR FILM BREAK-UP TIME













Analyses will be conducted as described in Section 14.2.1.



#### 15. Summary of Efficacy Analyses



#### 16. Safety Analyses

All safety analyses will be conducted using the safety population.

#### 16.1 Adverse Events

An AE is defined as any untoward medical occurrence associated with the use of an IP in humans, whether or not considered IP-related. An AE can be any unfavorable and unintended sign (e.g., an abnormal laboratory finding), symptom, or disease temporally associated with the use of an IP, without any judgment about causality. An AE can arise from any use of the IP (e.g., off-label use, use in combination with another drug or medical device) and from any route of administration, formulation, or dose, including an overdose. An AE can arise from any delivery, implantation, or use of a medical device, including medical device failure, subject characteristics that may impact medical device performance (e.g., anatomical limitations), and therapeutic parameters (e.g., energy applied, sizing, dose release, and anatomic fit) associated with medical device use. All AEs will be coded using the MedDRA 24.0.

Treatment-emergent adverse events (TEAE) are defined as any event that occurs or worsens on or after the first dose of randomized study drug.

Severity of an AE is defined as a qualitative assessment of the degree of intensity of an AE as determined by the Investigator or reported to him/her by the subject. The assessment of severity is made irrespective of relationship to study drug or seriousness of the event and should be evaluated according to the following scale:

- *Mild:* Event is noticeable to the subject, but is easily tolerated and does not interfere with the subject's daily activities.
- Moderate: Event is bothersome, possibly requiring additional therapy, and may interfere with the subject's daily activities.
- Severe: Event is intolerable, necessitates additional therapy or alteration of therapy, and interferes with the subject's daily activities.

The relationship of each AE to the IP should be determined by the investigator using these explanations:
### Protocol ST100-001 SAP, Version 1.0



- Definitely Related: Relationship exists when the AE follows a reasonable sequence from the time
  of IP administration, follows a known response pattern of the drug class, is confirmed by
  improvement on stopping the IP and no other reasonable cause exists.
- *Probably Related*: Relationship exists when the AE follows a reasonable sequence from the time of IP administration, follows a known response pattern of the drug class, is confirmed by improvement on stopping the IP and the suspect IP is the most likely of all causes.
- Possibly Related: Relationship exists when the AE follows a reasonable sequence from the time of IP administration, but could also have been produced by the subject's clinical state or by other drugs administered to the subject.
- *Unlikely to be Related*: Relationship uncertain to the investigational product. Likely to be related to factors other than investigational product but cannot be ruled out with certainty.
- Not Related: Concurrent illness, concurrent medication, or other known cause is clearly responsible
  for the AE, the administration of the IP and the occurrence of the AE are not reasonably related in
  time, or exposure to IP has not occurred.

TEAEs that are recorded as definitely related, probably related, and possibly related are considered as treatment-related TEAEs.

The expectedness of an AE should be determined based upon existing safety information about the IP using these explanations:

- Unexpected: An AE that is not listed in the Investigator's Brochure (IB) or is not listed at the specificity or severity that has been observed.
- Expected: An AE that is listed in the IB at the specificity and severity that has been observed.
- Not applicable: An AE unrelated to the IP.

All AEs that are mentioned in the IB as occurring with a class of products or as anticipated from the pharmacological/mechanical (or other) properties of the product but are not specifically mentioned as occurring with the particular product under investigation are to be considered unexpected

An overall summary will be presented that includes the number of events and the number and percentage of subjects who experienced at least one AE, ocular AE, and non-ocular AE by treatment group and over all subjects. This summary will also include the number of events and the number and percentage of subjects who experienced at least one TEAE, as well as breakdowns of TEAEs further categorized as ocular or non-ocular, TEAEs by severity, TEAEs by relationship to study drug, TEAEs causing premature treatment discontinuation, and SAEs. TE-SAEs will also be categorized as ocular or non-ocular, TE-SAEs by severity, TE-SAEs by relationship to study drug, TE-SAEs causing premature treatment discontinuation, and TE-SAEs leading to death.

Summaries will be provided for the following categories of AEs:

### Protocol ST100-001 SAP, Version 1.0



- Ocular and non-ocular TEAEs by SOC and PT
- Ocular and non-ocular TEAEs by SOC, PT, and maximal severity
- Ocular and non-ocular treatment-related TEAEs by SOC and PT
- Ocular and non-ocular TE-SAEs by SOC and PT
- Ocular and non-ocular TEAEs by SOC, PT and study day of onset (Day 8 or prior, After Day 8 to Day 15, and After Day 15 to Day 29).

If a subject reports the same PT multiple times within the same SOC, that PT will only be reported once within that SOC. As with the PT, if a subject reports multiple conditions within the same SOC, that SOC will only be reported once. In the summaries, SOCs and PTs within SOCs will be listed in order of descending frequency for all subjects.

All AEs for screened subjects, ocular AEs, non-ocular AEs, and SAEs for randomized subjects will be presented in subject listings.

# 16.3 Slit-Lamp Biomicroscopy Examination







### 16.5 Undilated Fundoscopy Examination



## 16.6 Urine Pregnancy Test



# 17. Interim Analyses

No interim analyses are planned.

## 18. Changes from Protocol-Stated Analyses

CFB-V2 Post as defined in section 9.3 of this SAP will be analyzed at Visit 3 (Day 2), Visit 4 (Day 4), Visit 5 (Day 8) Pre-CAE®, Visit 6 (Day 15) Pre-CAE®, and Visit 7 (Day 29) Pre-CAE®.

### 19. References

There are no applicable references for this SAP.

# 20. Revision History

Documentation of revision to the SAP will commence after approval of the final version 1.0.



# 21. Tables

Tables (10 tables total) that will be included in the topline delivery are shown in **boldface** font.

















23. Figures







24. Appendices











